CLINICAL TRIAL: NCT02819544
Title: Prospective, Two-center , Randomized, ITT , Parallel Group Evaluating the Interest of the Instillation of Saline Intraperitoneally (INSI ) Versus Instillation of Naropin the Surgical Site Versus Lung Recruitment Maneuvers ( PVM ) in the Management of Pain After Laparoscopic Cholecystectomy in Ambulatory Care
Brief Title: Evaluation of the Interest of the Instillation of Saline Intraperitoneally (INSI ) Versus Instillation of Naropin the Surgical Site Versus Lung Recruitment Maneuvers ( PVM ) in the Management of Pain After Laparoscopic Cholecystectomy in Ambulatory Care
Acronym: VSD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI2015_843_0020
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Surgery; Pain
Keywords: Digestive System
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Active Comparator): Ropivacaine 7.5 mg/mL administration
  Interventions: Drug: Ropivacaine administration
- Sodium chloride (Placebo Comparator): NaCl 0.9% administration
  Interventions: Drug: Sodium chloride administration

INTERVENTIONS:
Drug: Sodium chloride administration — Sodium chloride administration
  Arms: Sodium chloride
Drug: Ropivacaine administration — Ropivacaine administration
  Arms: Ropivacaine

SUMMARY:
Known to reduce analgesics and length of hospitalization in conventional surgery, laparoscopy is characterized by frequent post-operative pain and can decrease the patient's quality of immediate postoperative life and sometimes the results of decision ambulatory care.

In order to reduce these postoperative pain, various methods have been evaluated in numerous studies to determine their analgesic role.

As part of abdominal surgery, local anesthetics (Naropin (Ropivacaine)) are generally administered in the end of surgery to reduce postoperative pain and promote recovery of the patient. In addition, it is also possible to instill the anesthetic directly into the abdominal cavity reducing pain transmitted by nociceptor viscera.

In recent years, new methods have been proposed such as lung recruitment maneuvers and the instillation of saline solution to reduce postoperative pain.

However, no recommendation is on the use of intraperitoneal saline under the management of postoperative pain after laparoscopic cholecystectomy in ambulatory care.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 80 years
* Patients with biliary pathology requiring cholecystectomy
* Patients with signed consent
* Patient eligible to outpatient care
* No allergy to Naropin
* Support by laparoscopy
* Patients affiliated to a social security s

Exclusion Criteria:

* Contraindications for laparoscopy
* Contraindications to outpatient surgery
* Patients with an allergy to paracetamol or tramadol
* Patient with an addiction to painkillers and / or alcohol
* Patient with a disease causing chronic pain
* Patient using analgesics bearing 1 , 2 or 3 chronically
* Pregnant or breastfeeding women , of reproductive age without effective contraception
* Minor Patient,
* Contraindication to surgery,
* Physical or psychological state does not allow the patient's participation in the study ,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Pain measured by visual analog scale (VAS) | between first postoperative day and 6th postoperative day

SECONDARY OUTCOMES:
global pain measured by BPI (Brief Pain Inventory) scale | 30th postoperative day
analgesics use | 30th postoperative day
global morbidity | 30th postoperative day
specific complications for each treatment | 30th postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc REGIMBEAU, MD, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - CH Beauvais, Beauvais